CLINICAL TRIAL: NCT04121091
Title: Pramipexole Augmentation to Target Anhedonia in Depression - a Pilot Study
Brief Title: Pramipexole to Target "Anhedonic Depression"
Acronym: PILOT-PRAXOL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Daniel Lindqvist, Principal Investigator, Region Skane
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-001907-19
Record Dates: First submitted 2019-10-04; First posted 2019-10-09 (Actual); Results first posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-04

CONDITIONS: Depression, Bipolar; Depression, Unipolar; Dysthymia; Anhedonia
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder; Dysthymic Disorder; Anhedonia | interventions — Pramipexole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pramipexole (Experimental)
  Interventions: Drug: Pramipexole Pill

INTERVENTIONS:
Drug: Pramipexole Pill — Add-on pramipexole

SUMMARY:
The heterogeneity of depression suggests that different neurocircuits and pathophysiological mechanisms are involved. Anhedonia - the inability to experience pleasure from, or the lack of motivation to carry out, usually enjoyable activities - is an endophenotype within the depression spectrum, with a distinct pathophysiology of dopaminergic mesolimbic projections. Anhedonia is common in depression and associated with treatment resistance. Pramipexole, an agonist to the dopamine -receptor 3, is an established treatment of Parkinson's disease. Based on its mechanism of action, pramipexole might be efficacious in a subtype of depression characterized by anhedonia and lack of motivation - symptoms linked to dopaminergic hypofunction. In this proof-of-concept pilot study the investigators test the anti-anhedonic and antidepressant effects of add-on pramipexole using an "enriched population study design" including only depressed patients with significant anhedonia. To understand the neurobiology of anhedonia in depression and to identify treatment predictors, the investigators also do assessments of anhedonia-related neurocircuitry using (f)MRI and blood biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤75.
2. Diagnosis of unipolar depression; bipolar disorder in depressive phase or dysthymia.
3. Symptoms of depression; Total-score ≥ 18, measured by Montgomery-Åsberg Depression Rating Scale (MADRS).
4. Symptoms of anhedonia; Total-score < 27, measured by Dimensional Anhedonia Rating Scale (DARS).
5. Ongoing treatment with at least one antidepressant drug ≥ 4 weeks without major changes in dosage. Patients with bipolar disorder must have a mood-stabilizing drug treatment.
6. Must sign an informed consent. -

Exclusion Criteria:

1. Ongoing pregnancy, breastfeeding or planning for pregnancy.
2. High suicidality assessed by the researcher with medical degree.
3. Ongoing substance use disorder (last 12 month).
4. Diagnosis of psychosis.
5. Ongoing involuntary psychiatric treatment.
6. History of Impulse-control disorder or current ADHD diagnosis.
7. Diagnosis of Intellectual disability, dementia, or other circumstances leading to difficulties to understand the implications of participating in the study and to give informed consent.
8. Diagnosis of renal failure (eGFR < 50 ml/min/1,73 m2 ) or severe cardiovascular disease (defined as symptoms of heart failure NYHA class 2).
9. Recently committed to psychotherapy (during the last 6 weeks) or planning for psychotherapy during the participation of the study.
10. Ongoing ECT-treatment.
11. Other diseases, disorders or medical treatments that according to the researchers might influence the results of the study or increases the risks of the study. Such as Parkinson's disorder, liver failure, cancer not in remission (for at least over a year).
12. Confirmed or suspected allergy to the active substance or excipients of the drug used in this study.
13. Committed to other trials
14. Other reasons that according to the researcher might prevent the subject to fulfill the obligations of the study. For example insufficient drug compliance. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2021-03-18 (Actual); Study Completion 2021-03-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatry Clinic, Lund, Region Skåne, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from outpatient clinics in Lund, Sweden. All study visits were conducted via the adult psychiatric clinic in Lund, Baravägen 1, 221 85, Lund during the period 4 Oct 2019 - 18 Mar 2021.
Pre-assignment Details: 12 patients with unipolar or bipolar, moderate-to-severe, depression were assigned to active open-label treatment with pramipexole. The sample was enriched for significant anhedonia symptoms, enrolling only patients with a score of <27 on the Dimensional Anhedonia Rating Scale (DARS, inverse scale). 1 dropout pre-assignment/pre-treatment.
Groups:
- Pramipexole: Active treatment, open-label, with the dopamine agonist pramipexol individually titrated to highest tolerable dose (max 4,5 mg salt) daily. Administration: tablets orally.
Period: Overall Study
Arm/Group | Pramipexole
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Open-label, only one arm
Groups:
- Pramipexole: 12 patients
Arm/Group | Pramipexole
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  Sweden | 12
Tobacco users [Number; unit: Participants] | 5
hsCRP [Mean (Standard Deviation); unit: mg/L] — Serum high sensitivity C-reactive peptide
  mg/L | 3.8 (4.7)
Concurrent pharmacological treatment [Number; unit: Participants] — Ongoing psychoactive treatment at baseline
  Participants
    SSRI users | 5
    SNRI users | 6
    NDRI users | 2
    Antipsychotics users | 0
    Mood stabilizers users | 2
ECT [Count of Participants; unit: Participants] — Previously treated with electro-convulsive therapy
  Participants | 4
Anxiety comorbidity [Count of Participants; unit: Participants] — Anxiety disorder diagnosis at baseline
  Participants | 6
Number of previous antidepressants [Median (Full Range); unit: Number of different antidepressants] — Median number of previously tried antidepressant treatments
  Number of different antidepressants | 5 [2 to 14]

OUTCOME MEASURES:

1. Primary Outcome: Dimensional Anhedonia Rating Scale (DARS) Score
Description: Change in anhedonia symptoms (total score on the DARS). The range is 0-68, lower score indicating more severe anhedonia.
Time Frame: baseline to week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 12
score on a scale
  DARS total score baseline | 15.75 (6.440)
  DARS total score week 10 | 33.08 (11.782)

2. Secondary Outcome: Response
Description: Montgomery Åsberg Depression Rating Scale (MADRS). The range is 0-60, lower score indicating less general depressive symptoms.
  Response definition: reduction of at least 50% Remission definition: MADRS total score equal to or below 10
Time Frame: baseline to week 10
Measure: Count of Participants; unit: Participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 12
Participants
  Responders | 4
  Non-responders | 8

3. Secondary Outcome: Montgomery Åsberg Depression Rating Scale (MADRS) Score
Description: Change in depression symptoms (total score on the MADRS). The range is 0-60, lower score indicating less general depressive symptoms.
Time Frame: baseline to week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 12
score on a scale
  MADRS total score baseline | 26.33 (4.185)
  MADRS total score week 10 | 15.67 (6.401)

4. Secondary Outcome: Snaith-Hamilton Anhedonia Pleasure Scale
Description: Change in anhedonia symptoms (total score on the Snaith-Hamilton Anhedonia Pleasure Scale) score 0-1-2-3. Range 0-32. Higher score indicating more intense anhedonic symptoms.
Time Frame: baseline to week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 12
score on a scale
  SHAPS total score baseline | 30.00 (5.592)
  SHAPS total score week 10 | 17.50 (6.389)

5. Secondary Outcome: Generalized Anxiety Disorder-7
Description: Change in anxiety symptoms (total score on the the Generalized Anxiety Disorder-7 scale = GAD-7). Range 0-21. Higher score indicating more anxiety.
Time Frame: baseline to week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 12
score on a scale
  GAD-7 total score baseline | 9.64 (6.087)
  GAD-7 total score week 10 | 6.18 (6.570)

6. Secondary Outcome: Insomnia Severity Index
Description: Change in insomnia symptoms (total score on the the Insomnia Severity Index scale = ISI). Range 0-28. Higher score indicating more insomnia symptoms.
Time Frame: baseline to week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 11
score on a scale
  ISI total score baseline | 15.73 (6.182)
  ISI total score week 10 | 10.27 (4.839)

7. Secondary Outcome: Fatigue Severity Scale
Description: Change in fatigue symptoms (total score on the the Fatigue Severity scale = FSS). Range 9-63. Higher score indicating more fatigue.
Time Frame: baseline to week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 11
score on a scale
  FSS total score baseline | 46.45 (12.581)
  FSS total score week 10 | 38.45 (15.807)

8. Secondary Outcome: The Apathy Evaluation Scale
Description: Change in apathy symptoms (total score on the the The Apathy Evaluation Scale = AES). Range 0-54. Higher score indicating more severe apathy.
Time Frame: baseline to week 10
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pramipexole
Number analyzed (Participants) | 11
score on a scale
  AES total score baseline | 52.55 (6.905)
  AES total score week 10 | 36.18 (9.152)

9. Secondary Outcome: Change in Inflammatory Biomarkers
Description: The investigators will measure blood levels of Interleukin-6 (IL-6), C-reactive protein (CRP), Tumor Necrosis Factor Alpha (TNF), and White Blood Cell count (WBC) at baseline and at study completion. The investigators will test if baseline levels and treatment-associated change in inflammatory markers can predict treatment response
Time Frame: baseline to week 10
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pramipexole
Number analyzed (Participants) | 12
mg/L
  CRP at baseline | 3.8 (4.7)
  CRP at week 10 | 2.6 (3.5)

10. Secondary Outcome: Participation in fMRI With MID-task
Description: fMRI = functional magnetic resonance tomography. Structural imaging, followed by resting-state functional imaging, diffusion tensor imaging and thereafter the MID (monetary incentive delay) task.
Time Frame: baseline to week 10 (and baseline data as potential predictor)
Measure: Count of Participants; unit: Participants
Arm/Group | Pramipexole
Number analyzed (Participants) | 12
Participants
  Participating in fMRI | 8
  Not participating in fMRI | 4

ADVERSE EVENTS:
Time Frame: For each participant, adverse event data was collected for 14 weeks: every week for 10 weeks and an additional check-up at week 14.
Description: According to EU regulation 536/2014 (Clinical Trials Regulation, CTR).
Arm/Group | Pramipexole
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pramipexole (N=12)
Headache (General disorders) | 10
Nausea (General disorders) | 9
Fatigue (General disorders) | 3
Skin rashes (Skin and subcutaneous tissue disorders) | 3
Loss of appetite (Metabolism and nutrition disorders) | 2
Vertigo (General disorders) | 2
Depressed mood (Psychiatric disorders) | 1
Agitation (mild) (Psychiatric disorders) | 1
Overeating (Psychiatric disorders) | 1
Palpitations (Cardiac disorders) | 1
Mania (Psychiatric disorders) | 0

LIMITATIONS AND CAVEATS:
Inherent limitations and caveats of this test-of-feasibility study: small-scale (small sample) and open-label design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT04121091/Prot_SAP_000.pdf